CLINICAL TRIAL: NCT06913738
Title: A Pragmatic Non-randomized Controlled Study Evaluating the Efficacy of a Dimensional Adaptation of Good Psychiatric Management (GPM-extended) Compared to a Classic Outpatient Good Psychiatric Management Treatment for Patient Fulfilling Criteria for Borderline Personality Disorder
Brief Title: Evaluation of a Dimensional Adaptation of Good Psychiatric Management (GPM-extended) for the Treatment of Borderline Personality Disorder
Acronym: EPSYLIA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: AddiPsy (Other)
Collaborators: Clinique Caradoc (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-A00475-42
Record Dates: First submitted 2025-03-31; First posted 2025-04-06 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-03

CONDITIONS: Borderline Personality Disorder; Narcissism; Obsessive Compulsive Personality Disorder; Personality Disorder
Keywords: Personality disorder; borderline personality disorder; good psychiatric management; psychotherapy; dimensional
MeSH Terms: conditions — Borderline Personality Disorder; Compulsive Personality Disorder; Personality Disorders

STUDY DESIGN:
Intervention Model Description: The EPSYLIA study is a controlled, non-randomized, open-label trial using a "here-elsewhere" methodology (i.e., patient inclusion depends on the center to which each individual is referred).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- GPM-Extended group (ADDIPSY, Lyon, France) (Experimental): Participants receive a one-year outpatient treatment based on GPM-extended, a dimensional adaptation of Good Psychiatric Management for BPD. It includes weekly 1-hour individual therapy focused on dominant personality dilemmas (abandonment, self-esteem, control), guided by structured clinical and psychometric assessment. Psychiatric case management (30 min every 3 weeks) addresses medication and coordination of care. Group components include at least one 6-week psychoeducation program (borderline, narcissistic, or obsessive-compulsive focus) and, for high emotion dysregulation, an 18-week DBT skills training group.
  Interventions: Behavioral: GPM-Extended
- Classic GPM (Clinique CARADOC, Bayonne, France) (Active Comparator): Participants receive a one-year outpatient treatment based on classic Good Psychiatric Management (GPM) for BPD. It includes weekly 1-hour individual therapy focused on interpersonal hypersensitivity, delivered by a GPM-trained therapist. Psychiatric case management (30 min every 3 weeks) addresses medication and coordination of care. Group interventions include a 6-week psychoeducation group on BPD and, for patients with high emotion dysregulation, an 18-week DBT skills training group.
  Interventions: Behavioral: Classic GPM

INTERVENTIONS:
Behavioral: GPM-Extended — GPM-extended is a dimensional adaptation of Good Psychiatric Management (GPM) that retains its core principles-validation, real-life focus, alliance building-while enhancing flexibility and personalization. It emphasizes diagnostic clarity, treatment prioritization, and individualized psychoeducation based on three key personality dilemmas: fear of abandonment, self-esteem dysregulation, and control dependency. These dilemmas guide the focus of therapy and case management. Treatment goals are collaboratively set and regularly reassessed to align with the patient's evolving needs. The intervention includes weekly individual therapy and tailored group programs, with clinical strategies adapted to each dominant dilemma.
  Arms: GPM-Extended group (ADDIPSY, Lyon, France)
Behavioral: Classic GPM — The classic GPM group follows the validated and manualized version of Good Psychiatric Management (GPM) for BPD. It emphasizes symptom stabilization through weekly individual therapy and pragmatic case management every 3 weeks. Unlike GPM-extended, it uses a uniform therapeutic framework rather than tailoring treatment to individual personality dilemmas,.The intervention includes weekly individual therapy and standardized group programs, with clinical strategies applied uniformly across patients, centered on interpersonal hypersensitivity and building stable life roles.
  Arms: Classic GPM (Clinique CARADOC, Bayonne, France)

SUMMARY:
The goal of this clinical trial is to evaluate whether a dimensional adaptation of Good Psychiatric Management (called GPM-extended) is more effective than classic Good Psychiatric Management (GPM) in treating adult patients with borderline personality disorder (BPD). Briefly, the GPM-extended model integrates elements from existing adaptations of GPM for narcissistic and obsessive-compulsive personality disorders. It aims to provide a more personalized and dimensional approach to treatment, tailored to each patient's specific personality dysfunction and interpersonal triggers.

The main questions it aims to answer are:

* Does GPM-extended improve overall BPD symptom severity more than classic GPM after one year of treatment?
* Does GPM-extended lead to better outcomes in related clinical domains (e.g., personality functioning, emotional regulation, social functioning...) ?

Researchers will compare two groups:

* Patients treated in a center using the GPM-extended program.
* Patients treated in a center using the classic GPM program. In each group, patients will receive weekly outpatient psychiatric care for one year.

In terms of evaluation, patients will be evaluated at baseline, 4 months, 8 months, and 1 year. They will undergo both clinician-administered and self-report assessments to measure BPD symptoms and other relevant psychological dimensions.

This study hopes to contribute to the development of dimensional evidence-based treatments for personality disorders.

DETAILED DESCRIPTION:
Personality disorders (PD) are among the most common psychiatric disorders, the most studied being borderline personality disorder (BPD), a disorder that affects approximately 1.6% of the general population and is characterised by significant difficulties in emotion regulation, identity and interpersonal relationships. Currently, categories of PD are criticised and many authors have highlighted the need for a more dimensional assessment of PD, using the association of a general factor (described as the level of personality functioning, assessed on personal and interpersonal functioning) with several personality traits used to describe specific personality characteristics (negative affectivity, antagonism/dissociality, detachment, disinhibition, anankastia, psychoticism). The two main models are the DSM-5 alternative personality disorder model (AMPD) and the International Classification of Diseases 11th edition personality disorder model (ICD-11). In particular, several works have suggested that the BPD criteria are one of the most important markers of general personality functioning. While these new models offer new and very exciting possibilities in terms of diagnostic assessment, they have struggled to spread across clinical services ; and, to date, no evidence-based treatments have been developed from these models, limiting their usefulness. Furthermore, these models are also limited by the nature of personality traits (Criteria B), as these represent rigid and stable patterns of dysfunction that may be difficult to represent the complex day-to-day fluctuations in internal psychic coherence and interpersonal functioning characteristic of PD.

One of the most recent treatments for BPD is Good Psychiatric Management. This has proved as effective as specialist therapies such as dialectical behaviour therapy and has also been developed for other personality disorders (notably narcissistic and obsessional-compulsive PD). Each adaptation is based on a specific conceptualisation designed to represent the main ways in which an individual may dysfunction in the personal and interpersonal domains. According to these conceptualisations, each of these three personality disorders presents a specific trigger for its difficulties: threat to relational dependence with fear of rejection and abandonment for borderline PD, threat to self-esteem for narcissistic PD, threat to ability to control for obsessive PD. Thus, some authors have suggested that the development of an adaptation of the GPM incorporating both the central aspects of the dimensional models, but also each of these different triggers in a non-exclusive manner (as they may be found to a greater or lesser extent in each patient suffering from PD), could be both feasible and useful, in particular to resolve the above-mentioned problems.

Indeed, like traditional dimensional models, GPM offers the possibility of a dimensional approach, with personality functioning assessed by the presence or absence of the BPD criteria, and features of personal and interpersonal dysfunction considered holistically using GPM's trigger-based approach. However, unlike traditional dimensional models, GPM has been empirically tested and found to be effective in treating patients who meet the criteria for BPD. In addition, it offers an approach to personality characteristics that is simpler, easier to understand, more accessible to psychoeducation and closer to patients' everyday experience than the personality traits classically used in dimensional models. In addition, although each adaptation of the GPM focuses on different PDs, much of the content remains the same: making and announcing the diagnosis, psychoeducation, case management, recurrent assessment of progress and reassessment if there is no response, multimodal approach including psychodynamic and behavioural psychotherapy, anticipation of crises, and management of symptomatic medication, etc. This may be linked to the fact that, although each disorder has specific triggers/traits, the underlying level of personality functioning is represented by BPD criteria and is therefore expected to be treated by the same psychotherapeutic content. Thus, a dimensional adaptation of GPM seems both relevant and feasible to address the problems of conventional dimensional models, namely the lack of existence of evidence-based treatments associated with these models, and the aspecific nature of personality trait-based approaches.

Altogether, we developed a dimensional adaptation of the GPM (GPM-extended), aiming to treat patients fulfilling the criteria for BPD dimensionally by incorporating elements from the adaptations for narcissistic and obsessional personality disorders. In terms of content, GPM-extended takes the common part of the treatment from the three adaptations and uses it as a basis, while also offering the possibility of constructing treatment goals and exposure targets that are much more specific to a given patient, in particular by carrying out an initial assessment and prioritisation of the various triggers. If this adaptation were to be shown to be effective, it would ultimately improve the diagnostic assessment and management of patients fulfilling BPD criteria, by offering treatment that is more tailored to each profile.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years old)
* Diagnosis of borderline personality disorder according to the SCID-II (≥5 out of 9 criteria)
* Provision of written informed consent
* Affiliated with or beneficiary of the French national health insurance system

Exclusion criteria

* Age under 18 years
* Presence of a comorbid psychotic disorder, intellectual disability, severe antisocial traits, major substance use disorder incompatible with intensive therapy without abstinence, anorexia nervosa with somatic risk, or bipolar disorder in acute manic phase
* Individuals under legal protection (e.g., guardianship or legal safeguard)
* Individuals unable to cooperate or complete self- or clinician-administered questionnaires
* Individuals not affiliated with or not beneficiaries of the French national health insurance system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Estimated)
Dates: Start 2024-06-19 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Change in BPD symptom severity (ZAN-BPD total score) | From baseline to 1 year.
  Difference in mean change in total score on the Zanarini Rating Scale for Borderline Personality Disorder (ZAN-BPD), a clinician-rated instrument assessing the severity of borderline symptoms. Scores range from 0 to 36, with higher scores indicating greater severity of borderline symptoms.

SECONDARY OUTCOMES:
Change in BPD symptom dimensions (ZAN-BPD subscales) | From baseline to 1 year.
  Difference in mean change in ZAN-BPD subscale scores (affective, cognitive, impulsive, interpersonal), a clinician-rated instrument assessing the severity of borderline symptoms. The subscores assess subdimensions of borderline psychopathology, and range from 0 to 8 (for cognitive, impulsive, and interpersonal subscores), and from 0 to 12 (for affective subscore only). Higher scores indicating greater severity.
Change in personality functioning (LPFS-BF) | From baseline to 1 year.
  Change in total score and subscores (self and interpersonal functioning) on the Level of Personality Functioning Scale - Brief Form (LPFS-BF), a self-report tool assessing personality functioning impairment. Scores range from 12 to 48 (for total score), and from 6 to 24 (for both subscores). Higher scores indicates greater personality dysfunction.
Change in disability level (SDS) | From baseline to 1 year.
  Change in total and domain scores (work/school, social life, family life) on the Sheehan Disability Scale (SDS), a self-report measure of functional impairment. Scores range from 0 to 30 (for total score), and from 0 to 10 (for each subscore). Higher scores indicate greater disability.
Change in social functioning (QFS) | From baseline to 1 year.
  Change in frequency and satisfaction subscores on the Questionnaire de Fonctionnement Social (QFS), a self-report tool assessing social engagement and satisfaction. Scores range from 8 to 40 for both subscores. Higher scores indicate better social functioning.
Change in suicidal and self-harming behaviors (SBBDM-S) | From baseline to 1 year.
  Change in the number of self-reported suicide attempts and self-harming behaviors using the Suicidal Behavior and Body Damage & Modifications Scale (SBBDM-S), a self-report tool assessing lifetime prevalence and past number of suicidal behaviors and self-harming behaviors. There are no score ranges. The higher the score, the higher number of behaviors.
Change in self-reported BPD symptom severity (BSL-23) | From baseline to 1 year.
  Change in mean total score on the Borderline Symptom list 23 items, a self-report measure of borderline symptom severity. Scores range from 0 to 4. Higher scores indicate greater severity of borderline symptoms.
Change in narcissistic symptoms (PNI-B) | From baseline to 1 year.
  Change in grandiose and vulnerable subscores on the Pathological Narcissism Inventory - Brief Form (PNI-B), a self-report tool assessing both grandiose and vulnerable pathological narcissism. Both subscores range from 0 to 5. Higher scores indicate greater severity of narcissistic symptomatology.
Change in obsessive-compulsive personality traits (POPS) | From baseline to 1 year.
  Change in total score and subscores on the Pathological Obsessive-Compulsive Personality Scale (POPS), a self-report tool assessingobsessive-compulsive personality overall severity and specific traits, such as rigidity or perfectionism. Total score range from 49 to 294, and subscores range from 15 to 90 for rigidity, from 7 to 42 for emotional over-control, from 12 to 72 for maladaptive perfectionnism, and from 8 to 48 for reluctance to delegate and difficulty with change. Higher scores indicate greater severity of symptoms.
Change in impulsivity levels (UPPS) | From baseline to 1 year.
  Change in impulsivity scores using the original UPPS scale, a self-report tool assessing several dimensions of impulsivity (urgency, lack of premeditation, lack of perseverance, and sensation seeking). Scores range from 12 to 48 for urgency and sensation seeking, from 11 to 44 for premeditation, and from 10 to 40 for perseverance. Higher scores indicate greater impulsivity.
Change in emotion dysregulation (DERS) | From baseline to 1 year.
  Change in total score and subscores on the original version of the Difficulties in Emotion Regulation Scale (DERS), a self-report measure of emotional regulation difficulties. Scores range from 36 to 180 (for total scores), from 6 to 30 (for awareness, acceptance, impulse control subscores), from 5 to 25 (for clarity and engagement subscores), and from 8 to 40 for strategies subscore. Higher scores indicate greater emotion dysregulation.
Change in alexithymia (TAS-20) | From baseline to 1 year.
  Change in total score and subscores on the Toronto Alexithymia Scale - 20 items (TAS-20), a self-report tool assessing alexithymia (i.e., difficulty identifying and describing emotions). Total score ranges from 20 to 100, identification subscore ranges from 7 to 35, description subscore ranges from 5 to 25, and exterior-oriented thoughts subscore ranges from 8 to 40. Higher scores indicate greater severity of alexithymia.
Change in mentalizing abilities (MentS) | From baseline to 1 year.
  Change in total score and subscores on the Mentalization Scale (MentS), a self report tool assessing self-, other-mentalizing, and motivation to mentalize. Scores range from 28 to 140 (for total score), from 8 to 40 (for self-mentalizing), and from 10 to 50 (for other-mentalizing and motivation to mentalize). Higher score indicate better mentalizing abilities.
Change in attachment style (ECR-R) | From baseline to 1 year.
  Change in self-reported attachment anxiety and avoidance using the Experiences in Close Relationships-Revised (ECR-R) scale. Mean scores range from 1 to 7 for both subscores. Higher scores indicating higher attachment difficulties.
Change in entitlement beliefs (PES) | From baseline to 1 year.
  Change in score on the Psychological Entitlement Scale (PES), a self-report tool measuring entitlement (i.e., perceived deservingness and superiority). Score ranges from 9 to 56. Higher score indicates higher feelings of entitlement.
Change in defense mechanisms (DMRS-SR-30) | From baseline to 1 year.
  Change in defense mechanism patterns using the Defense Mechanism Rating Scale - Self Report (30 items). Score ranges from 0 to 112 for raw defense score (RDS), with each of the 28 individual defense scores, each of the seven defense level scores, each of the defensive category scores, and each of the defenseive factor scores expressed as a proportion of the RDS ranging from 0% to 100%. Moreover, the Overall Defensive Functioning score ranges from 1 to 7. Higher scores indicates higher use of defense mechanism.
Change in therapeutic alliance (WAI-SR) | From baseline to 1 year.
  Change in therapeutic alliance quality based on the Working Alliance Inventory - Self Report (WAI-SR), a self-report tool assessing therapeutic relationship using several dimensions (goal, task, and bond). Score ranges from 12 to 60 for total score, and from 4 to 20 for each subscore. Higher scores indicate better quality of the therapeutic relationship.
Change in personality traits (PID-5-BF) | From baseline to 1 year.
  Change in personality traits using the Personality Inventory for DSM-5 - Brief Form (PID-5-BF), a self-report tool assessing the five AMPD's maladaptive personality trait domains. Total score ranges from 0 to 75, each global subscore ranges from 0 to 15, and each mean subscore ranges from to 0 to 3. Higher scores indicate higher presence e of personality traits.
Change in the frequency of personality disorder diagnoses (SCID-II) | From baseline to 1 year.
  Comparison of the frequency of categorical personality disorder diagnoses using the SCID-II interview, an interviewer-rated diagnostic assessment of categorical personality disorders.
Change in the frequency of current psychiatric comorbidities (MINI) | From baseline to 1 year.
  Comparison of the frequency of psychiatric comorbidities assessed using the Mini International Neuropsychiatric Interview (MINI), an interviewer-rated diagnostic interview.
Partial, full treatment response, and remission rates (ZAN-BPD) | From baseline to 1 year.
  Rates of partial, full response, and remission based on change in ZAN-BPD scores, using criteria proposed by Ridolfi et al. (2019).
Dropout rate during treatment year | From baseline to 1 year.
  Number and percentage of participants who discontinued therapy before the end of the one-year program.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Blay, M.D., M.Sc, Principal Investigator — AddiPsy
Locations (2):
- France (2):
  - Clinique Caradoc, Bayonne
  - Addipsy, Lyon

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) used in published analyses will be shared through the Open Science Framework (OSF) platform for each resulting publication. This includes the datasets used in the statistical analyses and the corresponding statistical code. A separate protocol paper will be published prior to the main outcome publications. Data and code will be made available to promote transparency and open science, following the publication of each study output.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: The protocol paper will be published before the end of 2026. Other IPD and related materials will be made publicly available starting from the first publication of study results, for an indefinite period, to support transparency and open science.
Access Criteria: Access to data will be provided via a dedicated OSF link published alongside each article.

REFERENCES:
- [Background] Ridolfi ME, Rossi R, Occhialini G, Gunderson JG. A Clinical Trial of a Psychoeducation Group Intervention for Patients With Borderline Personality Disorder. J Clin Psychiatry. 2019 Dec 31;81(1):19m12753. doi: 10.4088/JCP.19m12753. PMID 31917907
- [Background] McMain SF, Guimond T, Streiner DL, Cardish RJ, Links PS. Dialectical behavior therapy compared with general psychiatric management for borderline personality disorder: clinical outcomes and functioning over a 2-year follow-up. Am J Psychiatry. 2012 Jun;169(6):650-61. doi: 10.1176/appi.ajp.2012.11091416. PMID 22581157
- [Background] McMain SF, Links PS, Gnam WH, Guimond T, Cardish RJ, Korman L, Streiner DL. A randomized trial of dialectical behavior therapy versus general psychiatric management for borderline personality disorder. Am J Psychiatry. 2009 Dec;166(12):1365-74. doi: 10.1176/appi.ajp.2009.09010039. Epub 2009 Sep 15. PMID 19755574
- [Background] Blay M, Benmakhlouf I, Duarte M, Perroud N, Greiner C, Charbon P, Choi-Kain L, Speranza M. Case reports: Using Good Psychiatric Management (GPM) conceptualizations in the dimensional assessment and treatment of personality disorders. Front Psychiatry. 2023 Jul 26;14:1186524. doi: 10.3389/fpsyt.2023.1186524. eCollection 2023. PMID 37564248
- [Background] Wright AGC, Ringwald WR, Hopwood CJ, Pincus AL. It's time to replace the personality disorders with the interpersonal disorders. Am Psychol. 2022 Dec;77(9):1085-1099. doi: 10.1037/amp0001087. PMID 36595407
- [Background] Wright AG, Hopwood CJ, Skodol AE, Morey LC. Longitudinal validation of general and specific structural features of personality pathology. J Abnorm Psychol. 2016 Nov;125(8):1120-1134. doi: 10.1037/abn0000165. PMID 27819472
- [Background] Sharp C, Wright AG, Fowler JC, Frueh BC, Allen JG, Oldham J, Clark LA. The structure of personality pathology: Both general ('g') and specific ('s') factors? J Abnorm Psychol. 2015 May;124(2):387-98. doi: 10.1037/abn0000033. Epub 2015 Mar 2. PMID 25730515
- [Background] Bach B, Kramer U, Doering S, di Giacomo E, Hutsebaut J, Kaera A, De Panfilis C, Schmahl C, Swales M, Taubner S, Renneberg B. The ICD-11 classification of personality disorders: a European perspective on challenges and opportunities. Borderline Personal Disord Emot Dysregul. 2022 Apr 1;9(1):12. doi: 10.1186/s40479-022-00182-0. PMID 35361271
- [Background] Hopwood CJ, Kotov R, Krueger RF, Watson D, Widiger TA, Althoff RR, Ansell EB, Bach B, Michael Bagby R, Blais MA, Bornovalova MA, Chmielewski M, Cicero DC, Conway C, De Clercq B, De Fruyt F, Docherty AR, Eaton NR, Edens JF, Forbes MK, Forbush KT, Hengartner MP, Ivanova MY, Leising D, John Livesley W, Lukowitsky MR, Lynam DR, Markon KE, Miller JD, Morey LC, Mullins-Sweatt SN, Hans Ormel J, Patrick CJ, Pincus AL, Ruggero C, Samuel DB, Sellbom M, Slade T, Tackett JL, Thomas KM, Trull TJ, Vachon DD, Waldman ID, Waszczuk MA, Waugh MH, Wright AGC, Yalch MM, Zald DH, Zimmermann J. The time has come for dimensional personality disorder diagnosis. Personal Ment Health. 2018 Feb;12(1):82-86. doi: 10.1002/pmh.1408. Epub 2017 Dec 11. No abstract available. PMID 29226598
- [Background] Gunderson JG, Herpertz SC, Skodol AE, Torgersen S, Zanarini MC. Borderline personality disorder. Nat Rev Dis Primers. 2018 May 24;4:18029. doi: 10.1038/nrdp.2018.29. PMID 29795363